CLINICAL TRIAL: NCT03926689
Title: Evaluating the Impact of Sending SMS Messages to Increase Egg Consumption Among Children One 1-2 Years of Age, a Cluster-randomized Controlled Trial in Kanchanpur, Nepal
Brief Title: SMS Messages to Increase Child Egg Consumption, a C-rct in Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helen Keller International (Other)
Collaborators: University of South Carolina (Other); University College, London (Other); International Food Policy Research Institute (Other); FHI 360 (Other); London School of Hygiene and Tropical Medicine (Other); United States Agency for International Development (USAID) (U.S. Federal Agency); Digital Broadcast Initiative Equal Access (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SIIegg2019-2020
Record Dates: First submitted 2019-03-08; First posted 2019-04-24 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: Dietary Habits
Keywords: egg consumption; dietary diversity; complementary feeding; South Asia; SMS
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Suaahara II Standard + SMS (Experimental): Suaahara II standard multi sectoral nutrition interventions (home visits, radio program, etc.) Suaahara II monthly SMS campaign targeting all adult household members of households in the 1000-day period between conception and a child's second birthday
  Interventions: Behavioral: SMS messages; Behavioral: Standard SII SBCC
- Suaahara II Standard (Active Comparator): Suaahara II standard multi sectoral nutrition interventions (home visits, radio program, etc.)
  Interventions: Behavioral: Standard SII SBCC

INTERVENTIONS:
Behavioral: SMS messages — A package of at least monthly SMS messages delivered to all adults in households with an individual in the 1000-day period between pregnancy and a child turning 2 years of age.
  Arms: Suaahara II Standard + SMS
Behavioral: Standard SII SBCC — Home visits/IPC; community events including food demo and key life events; and Bhanchhin Aama radio program episodes

SUMMARY:
Eggs are well-known to be a balanced source of protein, energy, fatty acids, and micronutrients and increasingly identified as an opportunity to improve nutrition of poor populations. Few implementation studies have been done globally, and none in South Asia, to assess the effectiveness of using behavior change programs to motivate households to increase egg consumption. Egg consumption is particularly poor in Nepal, but the government and development partners are implementing at scale policies and programs to address poor diets and other determinants of undernutrition, which is persistently high in Nepal.

This cluster-randomized controlled trial (c-RCT) aims to help address the gap in the evidence base regarding how to improve egg consumption. The c-RCT will evaluate the effectiveness of using short message service (SMS) messaging, layered into a large-scale behavior change program, to improve egg consumption and dietary diversity among children 1 to 2 years of age. A two-arm trial will be used to compare the following two strategies: 1) Suaahara II standard multi-sectoral nutrition interventions without any text messages and 2) Suaahara II standard multi sectoral nutrition interventions plus a SMS message campaign targeting all adult household members of households in the 1000-day period between conception and a child's second birthday.

DETAILED DESCRIPTION:
Eggs are well-known to be a balanced source of protein, energy, fatty acids, and micronutrients and increasingly identified as an opportunity to improve nutrition of poor populations. A recent trial in Ecuador showed dramatic improvements in child growth after consumption of eggs for only six months. This efficacy trial also showed that culturally appropriate strategies, taking local norms, values, and expectations into account, are important. Furthermore, small-scale egg production has proven to be an effective intervention to increase egg consumption among children. Few implementation studies have been done globally, and none in South Asia, to assess the effectiveness of using behavior change programs to motivate households to increase egg consumption.

Despite significant reductions in under-nutrition over the last several decades, Nepal persists as a nation with one of the highest prevalence of child undernutrition globally. There is substantial room for improvement in important nutrition-related behaviors, including poor diets. According to the 2016 Nepal Demographic and Health Survey (DHS), only about one-third of children 6 to 23 months of age receive a minimum acceptable diet, less than half (47%) eat foods from at least 4 of 7 food groups to attain minimum dietary diversity (DD), and not even 10% consume eggs. The Government of Nepal (GoN) and development partners have prioritized multi-sectoral (integrated) nutrition as a key development agenda. Suaahara II, a USAID-funded program (2016-2021), aims to reduce under-nutrition particularly among women and children in the 1000-day period between conception and a child's second birthday, a crucial window of opportunity during which interventions have optimal impact on child growth and development. Operational in 42 of Nepal's 77 districts, Suaahara II uses a district-wide approach and interventions cover nutrition, health, family planning, agriculture, governance, gender equality, and social inclusion.

Suaahara II's social and behavioral change communication (SBCC) interventions, using lessons learned from the first phase of Suaahara, prioritize 10 key behaviors for which knowledge-to-practice gaps persisted at the end of Suaahara I. Two of these 10 behaviors focus on dietary diversity: 1) mothers should eat a diverse diet, including eggs and meat, and 2) young children should eat a diverse diet, including eggs and meat. Suaahara II's SBCC approach includes a combination of interpersonal communication (IPC) (e.g., home visits for 1:1 counselling with Suaahara II frontline workers); community mobilization (e.g., health mothers group meetings; food demonstrations and key life event celebrations); mass media (i.e., an interactive weekly radio program known as Bhanchhin Aama); and as of 2018, a series of 35 SMS messages sent to 1000-day households (other than those residing in Kanchanpur, the trial district) to reinforce the promoted 10 key behaviors as well as regular contact with the health system.

The SMS messages started after monitoring data showed that over 95% of beneficiary households own a phone, including more than two-thirds of mothers. Each message is sent at a specific time to align with key times when a key nutrition-related health service contact point or important nutrition-related practice is needed during the 1000-day period (e.g., a reminder to go for antenatal care; an encouragement to continue exclusive breastfeeding for another two months when the child is 4 months). In pre-testing of this intervention in 2 districts with 1000-day mothers, Suaahara II found acceptability and interest to be high and a preference for text over voice messages as mothers noted that they can keep the former as record and messages were read when they had time providing them with flexibility; messaging could be as often as weekly; and mothers showed the messages to others and discussed about the content, even though not prompted to do so. The cost of sending SMS messages in Nepal is also lower than other behavior change methods which include costs for staff, travel, jobaids, and so on. For these reasons, SMS push-messaging has potential to be an effective tool for behavior change. Evidence of intervention effectiveness is lacking, however, and is particularly needed in Nepal where the Ministry of Health and Population is prioritizing the use of SMS push messages as part of their SBCC strategy for implementation of the Multi-sectoral Nutrition Plan.

While SMS messaging is promising, various mHealth, and more recently mNutrition, literature reviews have noted the lack of rigorous research designs to assess effectiveness of these interventions. Some mHealth studies have shown positive results; for example, in Zanzibar a trial showed that mobile messaging can improve antenatal care attendance. These studies are few, and mNutrition studies even fewer. To the investigator's knowledge, no studies have assessed the effectiveness of using mNutrition interventions to improve diets in South Asia. Recent formative research in Sri Lanka, however, suggests the potential effectiveness of using mobile phones to improve infant and young child feeding.

Growing mobile phone ownership in Nepal offers a potential mechanism for delivering nutrition messages to target groups in a time-saving and cost-effective way. While not everyone currently owns a phone, ownership is increasing even among quite remote populations. Given the combination of poor dietary diversity, limited reach of the health system, and having one of the fastest growing rates of mobile phone ownership among low- and middle-income countries, Nepal is an ideal setting for testing the use of SMS messages to promote ideal dietary practices.

This study aims to use the rigor of a randomized controlled trial (RCT) to address a gap in the evidence base regarding the effectiveness of using short message service (SMS) text messaging to improve dietary practices. The main research question is: are SMS messages, added to a large-scale behavior change program, an effective means of improving diets among children under 2 years of age? To assess the comparative effectiveness of delivering nutrition-related SMS messages, a two-arm trial will be used to compare the following two strategies: 1) Suaahara II standard multi-sectoral nutrition interventions, without any text messages, and 2) Suaahara II standard multi sectoral nutrition interventions plus a text message campaign targeting all adult household members of households in the 1000-day period between conception and a child's second birthday.

The c-RCT will involve a baseline survey in April/May 2019 and an endline survey in Nov-Jan 2021 (delayed due to covid-19, as originally planned data collection in April/May 2020 was not possible). The design is longitudinal at the cluster level but not at the household or individual level to be able to assess households with children aged 12-23 months at both baseline and endline. An SMS message intervention will begin in the trial district (Kanchanpur) only after data collection for the baseline has completed and will involve sending monthly text messages primarily about egg consumption and dietary diversity. About 4 months after the implementation starts, a mixed-methods process evaluation will be conducted to assess fidelity of program implementation and identify any challenges or bottlenecks to be addressed.

ELIGIBILITY:
Inclusion Criteria:

* household must have resided in the study cluster for the previous 12 months;
* household must have at least 1 child 12-23 completed months of age who was not acutely ill the previous day and does not have a disability preventing normal feeding; if a household has more than one child aged 12-23 months, but the children have different mothers, each mother is an eligible trial participant
* household must have at least one adult (18 years or older) residing in the household and owning a mobile phone
* household must be able and willing to register the phone number for the intervention and consent to inclusion in the survey for the trial.

Exclusion Criteria:

* a few clusters will be excluded from the study given their lack of representation of the overall study area (e.g., 2 clusters with less than 150 households which are all landless and without government resources; 1 cluster which is exclusively a Tamang population; and 1 cluster which is the main urban area)
* in the rare occurrence that in an eligible household, a mother has more than one child aged 12-23.9 months, then the youngest will be chosen in the trial and the other child excluded

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3301 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Child egg consumption | baseline and 12 months later
  Change in prevalence of any egg consumption in 24 hours prior to survey among children 12 to 23 months of age.
Child minimum dietary diversity | baseline and 12 months later
  Change in prevalence of obtaining minimum dietary diversity score (at least four of seven food groups) in previous 24 hours for children aged 12-23 months of age

SECONDARY OUTCOMES:
Child dietary diversity score | baseline and 12 months later
  Change in mean dietary diversity (range:0 lowest - 7 highest) in previous 24 hours for children 12 to 23 months of age
Adult caregiver egg consumption | baseline and 12 months later
  Change in prevalence of any egg consumption in previous 24 hours among adults residing in a household with a child 12 to 23 months of age
Adult minimum dietary diversity | baseline and 12 months later
  Change in prevalence of obtaining minimum dietary diversity score (at least five of ten food groups) in previous 24 hours among adults residing in a household with a child 12 to 23 months of age
Adult dietary diversity score | baseline and 12 months later
  Change in mean dietary diversity (range:0 lowest -10 highest) in previous 24 hours for adults residing in a household with a child 12 to 23 months of age
Infant and Young Child Feeding knowledge | baseline and 12 months later
  Change in mean knowledge score (range: 0-8) on core infant and young child feeding practices among adults residing in a household with a child 12 to 23 months of age
Health Mothers' Groups participation | baseline and 12 months later
  Change in prevalence of any participation in the last 3 months in a Female Community Health Volunteer-led group, by the mother of the survey child 12-23 months of age
Health Mothers' Groups participation frequency | baseline and 12 months later
  Change in number of times participated in the last 3 months in an Female Community Health Volunteer-led group by the mother of the survey child 12-23 months of age
Adult Bhanchhin Aama listenership | baseline and 12 months later
  Change in prevalence of any listenership in the last 3 months to Bhanchhin Aama, Suaahara II radio program, in the previous three months by any adult household member
Adult Bhanchhin Aama listenership frequency | baseline and 12 months later
  Change in number of times listened to Bhanchhin Aama, Suaahara II radio program, in the previous three months by any adult household member

CONTACTS AND LOCATIONS:
Overall Officials: Ed Frongillo, Principal Investigator — University of South Carolina; Aman Sen, Study Chair — Helen Keller International
Locations (1):
- Suaahara II/Helen Keller International, Nepal, Patan, Nepal

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Adhikari TB, Rijal A. E-mental health - An untapped opportunity in Nepal. Asian J Psychiatr. 2018 Dec;38:25-26. doi: 10.1016/j.ajp.2018.10.021. Epub 2018 Oct 23. No abstract available. PMID 30384225
- [Background] Barnett, I., Scott, N., Batchelor, S., Haddad, L., 2016. Dial "N" for nutrition? A Landscape Analysis of What We Know about m-Nutrition, m-Agriculture and m-Development.
- [Background] Campbell RK, Talegawkar SA, Christian P, LeClerq SC, Khatry SK, Wu LS, West KP Jr. Seasonal dietary intakes and socioeconomic status among women in the Terai of Nepal. J Health Popul Nutr. 2014 Jun;32(2):198-216. PMID 25076658
- [Background] Cunningham, K., Headey, D., Singh, A., Karmacharya, C., Rana, P.P., 2017. Maternal and Child Nutrition in Nepal: Examining drivers of progress from the mid-1990s to 2010s. Glob. Food Sec. 13, 30-37. https://doi.org/10.1016/j.gfs.2017.02.001
- [Background] Cunningham K, Singh A, Pandey Rana P, Brye L, Alayon S, Lapping K, Gautam B, Underwood C, Klemm RDW. Suaahara in Nepal: An at-scale, multi-sectoral nutrition program influences knowledge and practices while enhancing equity. Matern Child Nutr. 2017 Oct;13(4):e12415. doi: 10.1111/mcn.12415. Epub 2017 Jan 6. PMID 28058772
- [Background] Dulal B, Mundy G, Sawal R, Rana PP, Cunningham K. Homestead Food Production and Maternal and Child Dietary Diversity in Nepal: Variations in Association by Season and Agroecological Zone. Food Nutr Bull. 2017 Sep;38(3):338-353. doi: 10.1177/0379572117703264. Epub 2017 Apr 21. PMID 28429645
- [Background] Dumas SE, Lewis D, Travis AJ. Small-scale egg production centres increase children's egg consumption in rural Zambia. Matern Child Nutr. 2018 Oct;14 Suppl 3(Suppl 3):e12662. doi: 10.1111/mcn.12662. PMID 30332540
- [Background] FAO and FHI 360, 2016. Minimum Dietary Diversity for Women: A guide for measurement. http://www.fao.org/3/a-i5486e.pdf
- [Background] Gallegos-Riofrio CA, Waters WF, Salvador JM, Carrasco AM, Lutter CK, Stewart CP, Iannotti LL. The Lulun Project's social marketing strategy in a trial to introduce eggs during complementary feeding in Ecuador. Matern Child Nutr. 2018 Oct;14 Suppl 3(Suppl 3):e12700. doi: 10.1111/mcn.12700. PMID 30332535
- [Background] Houston, R., Shresha, M.B., Pomeroy, A., Wun, J., Sharma, I., 2014. Pathways To Better Nutrition Case Study: Nepal Strategic Background Report. Arlington, VA. https://www.popline.org/node/635850
- [Background] Lutter CK, Morris SS. Eggs: A high potential food for improving maternal and child nutrition. Matern Child Nutr. 2018 Oct;14 Suppl 3(Suppl 3):e12666. doi: 10.1111/mcn.12666. No abstract available. PMID 30332541
- [Background] Mildon, A., 2016. Use of Mobile Phone Technology to Support Improved Infant and Young Child Feeding Practices in Low-and Middle-income Countries: A Scoping Review. Univ. Toronto. University of Toronto. https://tspace.library.utoronto.ca/bitstream/.../Mildon_Alison_201611_MSc_thesis.pdf
- [Background] Ministry of Health 2017. Nepal Demographic and Health Survey 2016. Kathmandu.
- [Background] Morris SS, Beesabathuni K, Headey D. An egg for everyone: Pathways to universal access to one of nature's most nutritious foods. Matern Child Nutr. 2018 Oct;14 Suppl 3(Suppl 3):e12679. doi: 10.1111/mcn.12679. PMID 30332534
- [Background] Orton M, Agarwal S, Muhoza P, Vasudevan L, Vu A. Strengthening Delivery of Health Services Using Digital Devices. Glob Health Sci Pract. 2018 Oct 10;6(Suppl 1):S61-S71. doi: 10.9745/GHSP-D-18-00229. Print 2018 Oct 10. PMID 30305340
- [Background] Parajuli, J., Haynes, K.E., 2018. Cellular mobile telephony in Nepal. Lett. Spat. Resour. Sci. 11, 209-222. https://doi.org/10.1007/s12076-018-0212-7
- [Background] Singh A, Klemm RDW, Mundy G, Pandey Rana P, Pun B, Cunningham K. Improving maternal, infant and young child nutrition in Nepal via peer mobilization. Public Health Nutr. 2018 Mar;21(4):796-806. doi: 10.1017/S1368980017002993. Epub 2017 Nov 6. PMID 29103400
- [Background] Tilahun B, Smillie K, Bardosh KL, Murray M, Fitzgerald M, Cook V, Poureslami I, Forrest J, Lester R. Identifying Barriers and Facilitators of 13 mHealth Projects in North America and Africa: Protocol for a 5-Year Implementation Science Study. JMIR Res Protoc. 2018 Jul 3;7(7):e162. doi: 10.2196/resprot.9633. PMID 29970360
- [Background] World Health Organization, 2010. Indicators for assessing infant and young child feeding practices: part 1 definitions. Geneva.
- [Derived] Cunningham K, Cech S, Gupta AS, Rana PP, Humphries D, Frongillo EA. Text messages to improve young child diets: Results from a cluster-randomized controlled trial in Kanchanpur, Nepal. Matern Child Nutr. 2026 Mar;22(1):e13702. doi: 10.1111/mcn.13702. Epub 2024 Jul 17. PMID 39016667
- [Derived] Cunningham K, Pandey Rana P, Rahman MM, Sen Gupta A, Manandhar S, Frongillo EA. Text messages to improve child diets: Formative research findings and protocol of a randomised controlled trial in Nepal. Matern Child Nutr. 2023 Jul;19(3):e13490. doi: 10.1111/mcn.13490. Epub 2023 Mar 2. PMID 36864635